CLINICAL TRIAL: NCT05391347
Title: Effects of Orange Oil Aromatherapy on the Pain and Anxiety During Invasive Interventions in Patients With Hematopoietic Stem Cell Transplantation
Brief Title: Effects of Orange Oil Aromatherapy on the Pain and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Collaborators: Sinop University (Other); Acıbadem Atunizade Hospital (Other)
Responsible Party: Principal Investigator, DİLEK YILDIRIM, Assistant Prof., Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Orange oil aromatherapy
Record Dates: First submitted 2022-05-18; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Hematopoietic Transplantation; Bone Marrow Transplantation
Keywords: Hematopoietic stem cell transplantation; aromatherapy; pain; anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 3 ml of orange oil were dripping onto the sponge, and the patient was told to breathe slowly at a distance of 3 cm and to smell during the process
  Interventions: Other: Orange oil aromatherapy
- Control (No Intervention)

INTERVENTIONS:
Other: Orange oil aromatherapy — 5 minutes before the invasive procedure, 3 ml of orange oil were dripping onto the sponge, and the patient was told to breathe slowly at a distance of 3 cm and to smell during the process.
  Arms: Intervention

SUMMARY:
This randomized controlled experimental study was conducted prospectively with 80 patients with hematological malignancies were treated in the adult bone marrow transplant unit and adult hematology service of a private hospital between May 2021 and January 2022. Orange oil inhalation used in aromatherapy was applied to patients in the intervention group. Visual Analogue Scale and the State-Trait Anxiety Inventory used for data collection.

DETAILED DESCRIPTION:
Introduction: Invasive interventions such as peripheral intravenous cannula and port needle placement, and blood collection are often required for both inpatient and outpatient follow-up patients with hematological malignancies and hematopoietic stem cell transplantation patients. This long and difficult treatment process causes anxiety and emotional disorders in most patients. Although invasive initiatives in the treatment and monitoring process are widely implemented, they lead to pain, anxiety and discomfort, which is often ignored. This study conducted to assess the effect of orange oil inhalation used in aromatherapy on pain and anxiety levels in invasive interventions to treat patients with hematological malignancies and hematopoietic stem cells transplantation.

Methods: This randomized controlled experimental study was conducted prospectively with 80 patients with hematological malignancies were treated in the adult bone marrow transplant unit and adult hematology service of a private hospital between May 2021 and January 2022. Orange oil inhalation used in aromatherapy was applied to patients in the intervention group. Visual Analogue Scale and the State-Trait Anxiety Inventory used for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old,
* without communication problems,
* without allergy and respiratory system problems,
* who agreed to participate in the study

Exclusion Criteria:

* severe hypotension
* other allergic complications that made it difficult for patients to continue the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 5 minutes before the aromatherapy
  Visual Analog Scale; A scale applied on a straight line by marking a millimeter horizontal or vertical line. In this line, the 0 cm dot means "No Pain", while the 10 cm dot means "very bad pain". The patient marks the pain level on the scale. The marked point is measured using a tape measure and scored. Most studies so far show that visual analogue scale (VAS) is a reliable tool to use to assess the pain level
The State-Trait Anxiety Inventory (STAI) | 5 minutes before the aromatherapy
  In scale; there are 20 questions in the state area. It provides a four-point Likert type measurement. Scoring varies between 20-80. Although there is not a clear cut-off point, 39-40 points are often considered as the cut-off point of inventory. High score indicates high level of anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydin University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the researchers (i.e. upon rea-sonable request).